CLINICAL TRIAL: NCT05675046
Title: Multicenter Prospective Trial of Office-based Carpal Tunnel Release With Ultrasound Guidance (ROBUST)
Acronym: ROBUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonex Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90098-TP
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome; CTS
Keywords: Ultrasound Guided Carpal Tunnel Release; CTR-US; Office-Based; In Office; UltraGuideCTR
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Multicenter prospective single-arm trial of subjects with symptomatic Carpal Tunnel Syndrome treated with the Carpal tunnel Release with Ultrasound Guidance procedure using the UltraGuideCTR device in an office-based setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Carpal Tunnel Release with Ultrasound Guidance using the UltraGuideCTR device (Experimental): Participants who were treated with the Carpal Tunnel Release with Ultrasound Guidance procedure using the UltraGuideCTR device in the ROBUST Study.
  Interventions: Device: Carpal Tunnel Release with Ultrasound Guidance using the UltraGuideCTR device

INTERVENTIONS:
Device: Carpal Tunnel Release with Ultrasound Guidance using the UltraGuideCTR device — Participants who were treated with the Carpal Tunnel Release with Ultrasound Guidance procedure using the UltraGuideCTR device in the ROBUST Study.
  Other Names: UltraGuideCTR

SUMMARY:
Multicenter prospective single-arm trial of subjects with symptomatic Carpal Tunnel Syndrome treated with Ultrasound Guided Carpal Tunnel Release (CTR-US) in an office-based setting.

DETAILED DESCRIPTION:
Multicenter prospective single-arm trial of subjects with symptomatic Carpal Tunnel Syndrome treated with Ultrasound Guided Carpal Tunnel Release (CTR-US) in an office-based setting reporting the safety and effectiveness of office-based carpal tunnel release with ultrasound guidance (CTR-US) in patients with symptomatic carpal tunnel syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Clinical diagnosis of unilateral or bilateral idiopathic CTS
3. CTS-6 score >12 in target hand*
4. Median nerve cross-sectional area ≥10 mm2 in the proximal carpal tunnel region of the target hand measured by diagnostic ultrasound*
5. Prior failure of one or more nonsurgical treatment options (e.g., physical activity modification, bracing, splinting, corticosteroid injection)*
6. Subject agrees to complete follow-up questionnaires over a 24-month period
7. Subject has a valid smart phone number and/or email address to receive and answer follow-up questionnaires

Exclusion Criteria:

1. Prior surgery on the target wrist or hand with the exception of (a) trigger finger release or similar minor finger procedure (e.g., digital ganglion cyst removal, foreign body removal) that has clinically recovered, or release for DeQuervain's syndrome (1st dorsal compartment) that has clinically recovered*
2. History of prior surgical CTR in the target hand*
3. History of infection in the target hand*
4. History of prior surgery in the non-target hand, including CTR, within 3 months of enrollment or with persistent symptoms that interfere with normal daily activities or work at the time of consent
5. Planned surgical or interventional procedure on the contralateral hand within 3 months of the target hand procedure date*
6. Corticosteroid injection in the target hand within 6 weeks of study procedure date*
7. Presence of additional process in the target hand requiring additional intervention beyond carpal tunnel release (e.g. neurolysis, mass removal, tenosynovectomy)*
8. Clinically significant degenerative arthritis of the upper limb (shoulder to hand) on the target side*
9. Clinically significant inflammatory disease (including tenosynovitis) of the upper limb (shoulder to hand) on the target side*
10. Clinically significant trauma or deformity of the upper limb (shoulder to hand) on the target side*
11. Clinically significant vascular disease (including Raynaud's phenomenon) of the upper limb (shoulder to hand) on the target side*
12. Clinically significant neurological disorder (including complex regional pain syndrome) of the upper limb (shoulder to hand) on the target side*
13. Systemic inflammatory disease (e.g., rheumatoid arthritis, lupus)
14. Amyloidosis
15. Chronic renal insufficiency requiring dialysis
16. Diabetes not controlled by a stable dose of medication
17. Uncontrolled thyroid disease
18. Pregnant or planning pregnancy in the next 24 months
19. Workers' compensation subjects
20. Inability to provide a legally acceptable Informed Consent Form and/or comply with all follow-up requirements
21. Subject has other medical, social, or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations

Note: An asterisk (*) denotes that this criterion must be applied to the target hand for unilateral CTR-US procedures, or to both hands for simultaneous bilateral CTR-US procedures.

Clinically significant is defined as likely to interfere with the performance of the procedure in a safe and/or effective manner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2025-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Pistorio, MD, Principal Investigator — University of Nevada, Las Vegas
Locations (7):
- United States (7):
  - Orthopedic Associates, Fort Walton Beach, Florida
  - Vero Orthopaedics, Vero Beach, Florida
  - Georgia Hand, Shoulder & Elbow, Atlanta, Georgia
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - The Bone & Joint Surgery Clinic, Raleigh, North Carolina
  - New Braunfels Orthopaedic Surgery and Sports Medicine, New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: No
This study is privately funded and IPD will not be available for use beyond the study Sponsor or the participating Investigational Sites.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the ROBUST study began on February 16, 2023, and 149 subjects were enrolled. Enrollment was completed on June 30, 2023. Per the protocol, a subject was considered enrolled once they had signed the informed consent form, met all inclusion and exclusion criteria, and completed carpal tunnel release with Ultrasound guidance (CTR-US) using the UltraGuideCTR device.
Pre-assignment Details: Subjects could choose between having both hands treated (bilateral) at the same time if both hands met study criteria, or having one hand treated (unilateral) in the study. Bilateral patients with both hands treated are reported based on their averaged score, where applicable.
Period: Overall Study
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Started | 149
Completed | 149
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CTR-US: Participants who underwent Carpal Tunnel Release with Ultrasound Guidance (CTR-US) using the UltraGuideCTR device in the ROBUST Study.
Arm/Group | CTR-US
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 131
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 132
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Boston Carpal Tunnel Questionnaire - Symptom Severity Scale (BCTQ-SSS)
Description: The Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ-SSS) is a Carpal Tunnel Syndrome specific questionnaire that has been shown to be highly reproducible, internally consistent, valid, and responsive to clinical change in Carpal Tunnel Syndrome (CTS) and subject status post-carpal tunnel release (CTR). The BCTQ consists of 11 symptom severity questions (BCTQ-SSS). Scoring for the BCTQ- SSS ranges from 1 to 5, with higher scores indicating more severe symptoms, and is calculated as the mean of each response. The mean change score in BCTQ-SSS from baseline and 3-month follow-up are reported. Negative change scores indicate decreased symptom severity and positive change scores indicate increased symptom severity. Bilateral patients with both hands treated are reported based on their averaged score.
Time Frame: Baseline and 3 Months
Population: Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ-SSS) change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device: Participants who were treated with the Carpal Tunnel Release with Ultrasound Guidance procedure using the UltraGuideCTR device in the ROBUST Study. 146 out of 149 eligible participants completed the BCTQ-SSS at the 3-month visit and were analyzed for this endpoint. 3 participants did not complete the assessment.
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 146
units on a scale | -1.543 [-1.617 to -1.469]

2. Secondary Outcome: Time to Return To Normal Daily Activities (RTA)
Description: Time to return to normal daily activities will be defined as the number of days between treatment and the time the subject reports returning to normal daily activities, irrespective of work status.
Time Frame: 3 Months
Population: Time to return to normal daily activities
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 149
Days | 3.8 (6.66)

3. Secondary Outcome: Time to Return To Work Among Employed Subjects (RTW)
Description: Time to return to work will be defined as the number of days between treatment and the time the subject reports returning to work in any capacity.
Time Frame: 3 Months
Population: Time to return to work in days among employed subjects. 102/149 subjects were analyzed as only employed subjects were asked for return to work data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 102
Days | 7.0 (17.94)

4. Secondary Outcome: Boston Carpal Tunnel Questionnaire - Functional Status Scale (BCTQ-FSS)
Description: The Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ-FSS) additionally consists of 8 functional status questions. Scoring for the BCTQ-FSS ranges from 1 to 5, with higher scores indicating more functional limitation, and is calculated as the mean of each response. The mean change score in BCTQ-FSS from baseline to the 3-month follow-up are reported. Negative change scores indicate decreased functional limitation and positive change scores indicate increased functional limitation.
Time Frame: Baseline and 3 Months
Population: Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ-FSS) change at 3 months. 146 out of 149 eligible participants completed the BCTQ-FSS at the 3-month visit and were analyzed for this endpoint. 3 participants did not complete the assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 146
units on a scale | -0.969 [-1.055 to -0.882]

5. Secondary Outcome: Michigan Hand Questionnaire (MHQ)
Description: Michigan Hand Questionnaire (MHQ) is a validated, hand-specific questionnaire consisting of 37 questions in 6 domains:
  * Overall hand function
  * Activities of daily living
  * Work performance
  * Pain
  * Aesthetics
  * Satisfaction
  The total score ranges from 0 to 100. Higher scores indicate better hand performance; lower scores indicate lower hand performance. Mean change in the total MHQ score at the 3-month follow-up relative to baseline is reported.
Time Frame: Baseline and 3 Months
Population: Michigan Hand Questionnaire (MHQ) change at 3 months. 145 out of 149 eligible participants completed the MHQ at the 3-month visit and were analyzed for this endpoint. 4 participants did not complete the assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 145
units on a scale | 29.486 [27.443 to 31.528]

6. Secondary Outcome: Numeric Pain Scale
Description: The Numeric Pain Scale measures pain severity. Scoring for the Numeric Pain Scale ranges from 0 (indicating no pain) to 10 (indicating worst pain possible). The mean change scores in the Numeric Pain Scale from baseline and 3-month follow-up are reported. Negative change scores indicate decreased pain severity and positive change scores indicate increased pain severity. Bilateral patients with both hands treated are reported based on their averaged score.
Time Frame: Baseline and 3 Months
Population: Numeric Pain Scale change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 145
units on a scale | -3.472 [-3.706 to -3.237]

7. Secondary Outcome: EuroQoL 5-Dimension 5-Level (EQ-5D-5L)
Description: The EuroQol 5-Dimension 5-Level (EQ-5D-5L) is a generic preference-based questionnaire developed by the EuroQol Group to measure health-related quality of life. The EQ-5D-5L measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking consisting of: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Scoring for the EQ-5D-5L ranges from -0.57 (indicating lowest quality of life) to 1.00 (indicating highest quality of life). The mean change score in the EQ-5D-5L from baseline to the 3-month follow-up are reported. Negative change scores indicate decreased quality of life and positive change scores indicate increased quality of life.
Time Frame: Baseline and 3 Months
Population: EuroQol 5-Dimension 5-Level (EQ-5D-5L) change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 145
units on a scale | 0.138 [0.116 to 0.160]

8. Secondary Outcome: Number of Participants With Device and/or Procedure Related Adverse Events
Description: Participants with adverse events (AEs) occurring within 90 days of treatment and that are adjudicated as definitely related or probably related to the device or definitely related or probably related to the procedure will be included in this endpoint. The number of device- or procedure-related AEs within 90 days of treatment will represent an endpoint of the study.
Time Frame: 3 Months
Population: Participants with Procedure and/or Device-Related Adjudicated Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 149
Participants | 1

9. Secondary Outcome: Global Satisfaction
Description: Subjects were asked to rate their satisfaction with the carpal tunnel release procedure. The global satisfaction scale ranges from 1 to 5, with 1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Neither Satisfied nor Dissatisfied, 4 = Satisfied and 5 = Very Satisfied. The mean satisfaction score at the 3-month follow-up is reported. Bilateral patients with both hands treated are reported based on their averaged score. Higher scores indicate higher satisfaction; lower scores indicate lower satisfaction.
Time Frame: 3 Months
Population: Global satisfaction score at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device
Number analyzed (Participants) | 148
units on a scale | 4.4 (0.78)

ADVERSE EVENTS:
Time Frame: Adverse events were collected out to 1 year.
Description: AE could be reported 2 ways. 1) Documented by the site during the study procedure. 2) Subject reported an AE directly to the investigative site. If the site is notified of a potential AE by the subject, confirmation of the AE will occur by phone call with the subject or by asking the subject to return for a follow-up clinical evaluation.
Arm/Group | CTR-US
All-Cause Mortality (participants affected / at risk) | 0/149
Serious Adverse Events (participants affected / at risk) | 0/149
Other Adverse Events (participants affected / at risk) | 1/149
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTR-US (N=149)
Nerve Injury Median (non-digital) (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT05675046/Prot_SAP_000.pdf